CLINICAL TRIAL: NCT04408716
Title: Risk of Asymptomatic Cerebral Embolism During Atrial Fibrillation Ablation Using Smart Touch SF Catheter With Ablation Index Guided High-power Short-duration Strategy Versus Smart Touch Catheter With Standard Settings Evaluated by High-resolution Diffusion-weighted Magnetic Resonance Imaging Technique (REDUCE-IT Study)
Brief Title: Risk of Asymptomatic Cerebral Embolism During AF Ablation With AI-HPSD Strategy Versus Standard Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Professor, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REDUCE-IT Study
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Asymptomatic Cerebral Embolism; radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This study is a single center prospective single-blinded randomized controlled trial. Enrolled AF patients planning clinically-indicated catheter ablation is randomly assigned with 1:1 ratio to undergo catheter ablation with ablation index guided high-power short-duration strategy or the standard radiofrequency ablation technique. Besides the evaluation at baseline, all the participants will be followed up at 24-72 hours, 1 month and 3 months post ablation.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation Index Guided High-Power Short-Duration Group (Experimental): For patients assigned to undergo AF ablation with ablation index guided high-power short-duration strategy, point-by-point circumferential pulmonary vein ablation will be performed using the advanced STSF catheter under ablation index guided high power short duration strategy (Radiofrequency energy is set up at a power of 50 W, temperature of 43 °C, contact force of 5-20 gram, and flow rate of 20 mL/min; Target ablation index is set to 500 at the anterior wall and 350 at the posterior wall of left atrium).
  Interventions: Procedure: Ablation Index Guided High-Power Short-Duration Strategy
- Standard Radiofrequency Ablation Group (Active Comparator): For patients assigned to undergo AF ablation with standard radiofrequency ablation group, point-by-point circumferential pulmonary vein ablation will be performed using the ST catheter under standard radiofrequency ablation settings (Radiofrequency energy is set up at a power of 30 to 35 W, temperature of 43 °C, contact force of 5-20 gram, and flow rate of 17 to 30 mL/min. Target ablation index is set to 500 at the anterior wall and 350 at the posterior wall of left atrium).
  Interventions: Procedure: Standard Radiofrequency Ablation Technique

INTERVENTIONS:
Procedure: Ablation Index Guided High-Power Short-Duration Strategy — Point-by-point circumferential pulmonary vein ablation will be performed using the advanced STSF catheter under ablation index guided high power short duration strategy (Radiofrequency energy is set up at a power of 50 W, temperature of 43 °C, contact force of 5-20 gram, and flow rate of 20 mL/min; Target ablation index is set to 500 at the anterior wall and 350 at the posterior wall of left atrium).
  Arms: Ablation Index Guided High-Power Short-Duration Group
Procedure: Standard Radiofrequency Ablation Technique — Point-by-point circumferential pulmonary vein ablation will be performed using the ST catheter under standard radiofrequency ablation settings (Radiofrequency energy is set up at a power of 30 to 35 W, temperature of 43 °C, contact force of 5-20 gram, and flow rate of 17 to 30 mL/min. Target ablation index is set to 500 at the anterior wall and 350 at the posterior wall of left atrium).
  Arms: Standard Radiofrequency Ablation Group

SUMMARY:
The purpose of this prospective randomized controlled study is to evaluate the risk of asymptomatic cerebral embolism during catheter ablation of atrial fibrillation (AF) with AI-HPSD strategy versus standard radiofrequency ablation settings, with the diagnosis of asymptomatic cerebral embolism is determined by brain high-resolution diffusion-weighted magnetic resonance imaging technique.

DETAILED DESCRIPTION:
Radiofrequency catheter ablation is increasingly performed in patients with paroxysmal and persistent atrial fibrillation (AF) in recent decade. However, catheter ablation of AF is associated with the occurrence of procedure-related thromboembolic events, especially the risk of asymptomatic cerebral embolism detected by brain high-resolution diffusion-weighted magnetic resonance imaging (hDWI). Meanwhile, ablation index guided high-power short-duration (AI-HPSD) strategy with the advanced SmartTouch SurroundFlow (STSF) catheter is an increasingly used technique for catheter ablation of AF, which is proposed to be associated with relatively wider and superficial lesions, less risk of esophageal injury, and shorter procedure time plus higher rate of first-pass pulmonary vein isolation. Moreover, the advanced STSF catheter in AI-HPSD strategy features with the Surround Flow entire tip irrigation system, which is a wide-spread distribution of the irrigating solution (56 irrigation holes), resulting in homogenous cooling and protection from thrombus formation and reduced incidence of steam pops. Thus, comparing with the standard radiofrequency ablation technique using the SmartTouch (ST) catheter, the AI-HPSD strategy may associate with much lower risk of periprocedural asymptomatic cerebral embolism, with the application of advanced STSF catheter and shorter procedure time. Therefore, this study is designed as a prospective randomized controlled study to evaluate the risk of asymptomatic cerebral embolism during catheter ablation of AF with AI-HPSD strategy versus standard radiofrequency ablation settings, with the diagnosis of asymptomatic cerebral embolism is determined by brain hDWI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients≥18 years of age prior to obtaining the written informed consent.
2. Patients with electrocardiographically documented, symptomatic atrial fibrillation.
3. Patients is scheduled to undergo circumferential pulmonary vein antrum radiofrequency ablation.
4. Patient or patient's legal representative is able and willing to give informed consent.

Exclusion Criteria:

1. Moderate to severe valvular heart disease.
2. Contraindication for anticoagulation therapy.
3. Contraindication for Diffusion-Weighted MRI.
4. Ischemic stroke or transient ischemic attack within 6 months prior to the consent date.
5. Acute coronary syndrome within 3 months prior to the consent date.
6. Prior left atrial appendage occlusion device.
7. Prior septal occlusion device.
8. Left atrial size greater than 55 mm.
9. Conditions that prevent patient's participation in neurocognitive assessment (at physician's discretion).
10. Female patients who are pregnant or breast feeding or plan a pregnancy during the course of the study.
11. Simultaneous participation in another study.
12. Unwilling or unable to comply fully with the study procedures and follow-up requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of new asymptomatic cerebral embolic lesions determined by hDWI. | Within 3 days prior to the ablation；24-72 hours after AF catheter ablation procedure.
  The brain hDWI should be performed within 3 days prior to the ablation procedure to investigate previous cerebral lesions and reevaluated within 24-72 hours post ablation to determine the occurrence of new asymptomatic cerebral embolic lesions. The acute cerebral embolic lesion is typically defined as a new focal hyper-intense area detected on the diffusion-weighted sequence, and a hyper-intense signal intensity in the fluid-attenuated inversion recovery sequence, and meantime confirmed by apparent diffusion coefficient mapping as corresponding area of restricted diffusion to rule out a shine-through artifact.

SECONDARY OUTCOMES:
Cognitive functional status evaluated using the Montreal Cognitive Assessment (MoCA) test. | On the 1 day before and 24-72 hours and 3 months after the catheter ablation procedure.
  The Montreal Cognitive Assessment (MoCA) is known as a brief cognitive screening tool with a high sensitivity and specificity for detecting a mild cognitive impairment. All enrolled patients undergo a prospective assessment of their cognitive function using the MoCA test at 1 day before and 24-72 hours and 3 months after the catheter ablation procedure.
Overall complication rate during catheter ablation and up to 3 months follow up. | 3 months after the catheter ablation procedure.
  Overall complication rate after catheter ablation of AF.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affilliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt B, Szeplaki G, Merkely B, Kautzner J, van Driel V, Bourier F, Kuniss M, Bulava A, Nolker G, Khan M, Lewalter T, Klein N, Wenzel B, Chun JK, Shah D. Silent cerebral lesions and cognitive function after pulmonary vein isolation with an irrigated gold-tip catheter: REDUCE-TE Pilot study. J Cardiovasc Electrophysiol. 2019 Jun;30(6):877-885. doi: 10.1111/jce.13902. Epub 2019 Mar 25. PMID 30848001
- [Background] Yu Y, Wang X, Li X, Zhou X, Liao S, Yang W, Yu J, Zhang F, Ju W, Chen H, Yang G, Li M, Gu K, Tang L, Xu Y, Chan JY, Kojodjojo P, Cao K, Fan J, Yang B, Chen M. Higher Incidence of Asymptomatic Cerebral Emboli After Atrial Fibrillation Ablation Found With High-Resolution Diffusion-Weighted Magnetic Resonance Imaging. Circ Arrhythm Electrophysiol. 2020 Jan;13(1):e007548. doi: 10.1161/CIRCEP.119.007548. Epub 2020 Jan 14. PMID 31937118
- [Background] Providencia R, Albenque JP, Boveda S. The unfinished issue of ischaemic stroke and embolic events during catheter ablation of atrial fibrillation. Europace. 2017 May 1;19(5):881. doi: 10.1093/europace/euw027. No abstract available. PMID 28340141
- [Background] Yamane T. Silent Cerebral Embolism After Catheter Ablation for Atrial Fibrillation - Unresolved Issue or Too Much Concern? Circ J. 2016;80(4):814-5. doi: 10.1253/circj.CJ-16-0186. Epub 2016 Mar 7. No abstract available. PMID 26948985
- [Background] Kyriakopoulou M, Wielandts JY, Strisciuglio T, El Haddad M, Pooter J, Almorad A, Hilfiker G, Phlips T, Unger P, Lycke M, Vandekerckhove Y, Tavernier R, Duytschaever M, Knecht S. Evaluation of higher power delivery during RF pulmonary vein isolation using optimized and contiguous lesions. J Cardiovasc Electrophysiol. 2020 May;31(5):1091-1098. doi: 10.1111/jce.14438. Epub 2020 Mar 18. PMID 32147899
- [Background] Castrejon-Castrejon S, Martinez Cossiani M, Ortega Molina M, Escobar C, Froilan Torres C, Gonzalo Bada N, Diaz de la Torre M, Suarez Parga JM, Lopez Sendon JL, Merino JL. Feasibility and safety of pulmonary vein isolation by high-power short-duration radiofrequency application: short-term results of the POWER-FAST PILOT study. J Interv Card Electrophysiol. 2020 Jan;57(1):57-65. doi: 10.1007/s10840-019-00645-5. Epub 2019 Nov 12. PMID 31713704
- [Background] Okamatsu H, Koyama J, Sakai Y, Negishi K, Hayashi K, Tsurugi T, Tanaka Y, Nakao K, Sakamoto T, Okumura K. High-power application is associated with shorter procedure time and higher rate of first-pass pulmonary vein isolation in ablation index-guided atrial fibrillation ablation. J Cardiovasc Electrophysiol. 2019 Dec;30(12):2751-2758. doi: 10.1111/jce.14223. Epub 2019 Oct 21. PMID 31600006
- [Background] Chen S, Schmidt B, Bordignon S, Urbanek L, Tohoku S, Bologna F, Angelkov L, Garvanski I, Tsianakas N, Konstantinou A, Trolese L, Weise F, Perrotta L, Chun KRJ. Ablation index-guided 50 W ablation for pulmonary vein isolation in patients with atrial fibrillation: Procedural data, lesion analysis, and initial results from the FAFA AI High Power Study. J Cardiovasc Electrophysiol. 2019 Dec;30(12):2724-2731. doi: 10.1111/jce.14219. Epub 2019 Oct 13. PMID 31588620
- [Derived] Chen WJ, Gan CX, Cai YW, Liu YY, Xiao PL, Zou LL, Xiong QS, Qin F, Tao XX, Li R, Du HA, Liu ZZ, Yin YH, Ling ZY. Impact of high-power short-duration atrial fibrillation ablation technique on the incidence of silent cerebral embolism: a prospective randomized controlled study. BMC Med. 2023 Nov 23;21(1):461. doi: 10.1186/s12916-023-03180-3. PMID 37996906
- See also: Publications regarding the results of this Reduce-It Study. — https://bmcmedicine.biomedcentral.com/articles/10.1186/s12916-023-03180-3